CLINICAL TRIAL: NCT04509258
Title: Comparative Effectiveness of N-acetyl Cysteine, Acetyl L- Carnitine and Medicated Paraffin Oil in Acute Aluminium Phosphide Poisoning: A Clinical Trial
Brief Title: Effectiveness of N-acetyl Cysteine, Acetyl L- Carnitine and Medicated Paraffin Oil in Aluminium Phosphide Poisoning
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dalia K. Zaafar, lecturer of pharmacology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R 66/2019
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: the Study Focus to Improve the Standard of Care Used for Aluminuim Phosphide Poisoning and to Save Patients With the Minimal Organ Damage
Keywords: N-acetyl cysteine; Acety L- carnitine; paraffin oil; aluminium phosphide
MeSH Terms: interventions — Acetylcysteine; Acetylcarnitine; Ondansetron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- control group (Placebo Comparator): this group will have the standard and routine therapy of treatment of acute Aluminium Phosphide poisoning immediately after admission according to PCCA guidelines
  Interventions: Drug: Sodium Bicarbonate Powder and ondansetron
- N- acetyl cysteine grouo (Active Comparator): N-acetyl cysteine will be given at dose of 300mg/kg/d IV in the first day then 150 mg/kg/d IV in addition to standard of care according to PCCA guidelines
  Interventions: Drug: N-acetyl cysteine; Drug: Sodium Bicarbonate Powder and ondansetron
- Acetyl L-carnitine group (Active Comparator): Acetyl L-carnitine will be given at dose of 50 mg/kg IV once to be followed by additional doses of 15 mg/kg IV q4hr infused over 30 min. standard of care according to PCCA guidelines will also be provided
  Interventions: Dietary Supplement: acetyl L-carnitine; Drug: Sodium Bicarbonate Powder and ondansetron
- Medicated paraffin oil group (Active Comparator): Gastric decontamination with sodium bicarbonate (NaHCO3; 44 mEq, orally) and medicated paraffin oil (200 mL) will be administered in addition to standard of care according to PCCA guidelines
  Interventions: Drug: medicated paraffin oil; Drug: Sodium Bicarbonate Powder and ondansetron

INTERVENTIONS:
Drug: N-acetyl cysteine — a drug which can have an off label use as an antidot for aluminium phosphide poisoning in addition to sodium bicarbonate and ondansetron as standard of care
  Arms: N- acetyl cysteine grouo
Dietary Supplement: acetyl L-carnitine — Naturallu occuring amino acid derivative which can be taken as a dietary supplement involves in mitochondrial function and energy production and is suggested to have a role in lowering organ damage resulting from aluminium phosphide poisonong in addition to sodium bicarbonate and ondansetron as standard of care
  Arms: Acetyl L-carnitine group
Drug: medicated paraffin oil — refined mixture of liquid hydrocarbons which used as laxative and is suggested to reduce absorption of aluminium phosphide if taken within two hours of administration of the toxin in addition to sodium bicarbonate and ondansetron as standard of care
  Arms: Medicated paraffin oil group
Drug: Sodium Bicarbonate Powder and ondansetron — standard of care for treatment of aluminuim phosphide is provided for patients poisoned with aluminuim phosphide

SUMMARY:
Aluminium Phosphide is a pesticide used in developing countries to prevent rodents and pests from spoiling the harvested grains. it is presented as tablets which can be administered accidently to humans or for committing suicide. this pesticide is fatal even in small concentration as mortality rate can reach 75- 100% of cases. in this study researchers tried to add some supplements to the routine treatment to improve and decrease the fatality rate.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with history of acute intoxication with AlP presented to the Poison Control Center of Ain-Shams University hospitals during the period of the study

Exclusion Criteria:

1. Patients less than 18
2. Patients presented with delay time exceeding 12 hours after acute intoxication.
3. Patients with history of cardiac, renal or hepatic diseases.
4. Patients who show hypersensitivity to NAC, ALCAR or paraffin oil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
mortality rate reduction | 1 year
  the primary end point is to lower the mortality rate for patients poisoned with aluminium phosphide pellets
organ damage reduction | 1 year
  another primary end point is to reduce organ damage and injury for survivors

CONTACTS AND LOCATIONS:
Locations (1):
- Poison Control Center of Ain-Shams University hospitals, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: No
individual paticipant data is decided not to be shared for the privacy of the patients as patients in each group will be coded in numbers instead of their names